CLINICAL TRIAL: NCT04510077
Title: Study of SmartQuit, a Smartphone-Based Smoking Cessation Program
Brief Title: SmartQuit Program for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Life Sciences Discovery Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1001139; NCI-2020-05658 (Registry Identifier: NCI / CTRP); 8287 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2020-08-06; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Cigarette Smoking-Related Carcinoma; Tobacco-Related Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (SmartQuit) (Experimental): Patients use the SmartQuit program to learn and practice skill modules as often as they wish over 6 months.
  Interventions: Behavioral: SmartQuit Smoking and Tobacco Cessation Program; Other: Survey Administration

INTERVENTIONS:
Behavioral: SmartQuit Smoking and Tobacco Cessation Program — Use SmartQuit program
  Other Names: 2Morrow; SmartQuit
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial investigates how well a smartphone-based smoking cessation program called SmartQuit works to help patients stop smoking. SmartQuit is an smartphone application-based smoking cessation program that includes a defined program consisting of interactive evidence-based exercises for dealing more effectively with urges to smoke, a place to track desired behaviors, personalized plans for quitting, and a certificate of completion once the recommended program components are completed. SmartQuit may help patients quit smoking, lower healthcare costs and reduce premature tobacco-related deaths.

DETAILED DESCRIPTION:
OUTLINE:

Patients use the SmartQuit program to learn and practice skill modules as often as they wish over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Smokes at least five cigarettes daily for at least past 12 months
* Wants to quit in the next 30 days
* Interested in learning skills to quit smoking
* Resides in United States (US)
* Has at least daily access to their own smartphone
* Knows how to login and download a smartphone application from their smartphone
* Willing and able to read in English
* Not participating in other smoking cessation interventions (including our other intervention studies)
* Must be an employee of a company who is participating in recruitment
* Willing to complete one follow-up survey
* Provide email, phone, and mailing address

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-08-11 (Actual)

PRIMARY OUTCOMES:
Number of participants with 7-day cigarette smoking cessation at 2 months. | At 2 month follow-up
  No smoking at all in the past 7 or more days (7-day point prevalence quit rate).

SECONDARY OUTCOMES:
24-hour point prevalence quit rate | At 2 month follow-up
Change in number of cigarettes smoked per day | At 2 month follow-up
Number of intentional 24-hour quit attempts | At 2 month follow-up
Change in readiness to quit | At 2 month follow-up
  Differences in a participant's readiness to quit will be assessed by comparing their responses to the baseline survey readiness to quit questions with their responses to the 2 month follow-up survey
Nicotine dependence level | At 2 month follow-up
  Participants will share their nicotine dependence level via survey at their 2 month follow-up
Number of times logged into the application | At 2 month follow-up
  Will be assessed via 2 month follow-up survey
Time spent on the application | At 2 month follow-up
  Will be assessed via 2 month follow-up survey
Participant satisfaction with the application | At 2 month follow-up
  Will be assessed via 2 month follow-up survey
Participant opinion of the usefulness of the application for quitting smoking | At 2 month follow-up
  Will be assessed via 2 month follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Bricker, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No